CLINICAL TRIAL: NCT05567666
Title: A Real-word, Clinical Study to Evaluate the Performance of the Optilume® BPH Catheter System in Men With Symptomatic Benign Prostatic Hyperplasia (BPH)
Brief Title: Optilume BPH Catheter System in Benign Prostatic Hyperplasia (BPH)
Acronym: SUMMIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dean Elterman (Other)
Collaborators: Urotronic Inc. (Industry)
Responsible Party: Sponsor-Investigator, Dean Elterman, Lead Principal Investigator, Can-Am HIFU Inc.
Organization: Can-Am HIFU Inc. (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUMMIT (Protocol no.: 1001)
Record Dates: First submitted 2022-09-29; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Optilume; MIST
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: Optilume Catheter System, which is a Dilation Drug Coated Balloon (DCB) Catheter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental): Optilume Catheter System
  Interventions: Device: Optilume Catheter System

INTERVENTIONS:
Device: Optilume Catheter System — Optilume Catheter System, which is a Dilation Drug Coated Balloon (DCB) Catheter

SUMMARY:
A post-marketing study using Optilume Catheter System for benign prostatic hyperplasia.

DETAILED DESCRIPTION:
This is a post-marketing study for using Optilume Catheter System, which is a Dilation Drug Coated Balloon (DCB) Catheter, to treat benign prostatic hyperplasia. Participants will go through screening process which include uroflow test (measure the strength of urine flow), post-void residual volume by bladder scan, questionnaires and transrectal ultrasound (TRUS) to determine the eligibility to the study. Participants will be followed up for 1 year after Optilume treatment procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Male subject with symptomatic BPH NOTE: Symptomatic BPH is defined as an International Prostate Symptom Score (IPSS) ≥ 13 and peak urinary flow rate (Qmax) of ≤15 mL/sec
2. Prostate dimensions suitable for treatment with the Optilume BPH Catheter System in accordance with the approved Instructions for Use NOTE: Prostate volume between 20 to 80 gm and prostatic urethral length between 32 mm and 55 mm as determined by TRUS
3. Able to complete the study protocol in the opinion of the investigator

Exclusion Criteria:

1. Unable or unwilling to sign the Informed Consent Form (ICF) and/or comply with follow-up requirements
2. Unwilling to abstain from sexual intercourse or use a condom for 30 days post-procedure and a highly effective contraceptive for at least 6 months post-procedure
3. Presence of an artificial urinary sphincter or stent(s) in the urethra or prostate
4. Any prior minimally invasive intervention (e.g. TUNA, Balloon, Microwave, Rezūm, UroLift) or surgical intervention of the prostate
5. Confirmed or suspected malignancy of prostate or bladder
6. Active urinary tract infection (UTI) confirmed by culture
7. History of overt urinary incontinence requiring use of pads NOTE: Pad usage for post-micturition dribble is acceptable
8. Presence of confounding diagnoses impacting lower urinary tract symptoms or bladder function (e.g. urethral strictures, bladder neck contracture, neurogenic bladder, detrusor instability, bladder stones, etc.)
9. History of chronic urinary retention (e.g. PVR ≥300mL on two separate occasions, or catheter dependent drainage)
10. Anatomy (e.g. presence of false passage or size of meatus) is not suitable for treatment with the Optilume BPH Catheter System
11. Significant obstruction from median lobe in the opinion of the investigator
12. Disease or other health condition that is not suitable for this study

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 30 (Estimated)
Dates: Start 2022-11-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Responder Rate at 12 months | 12 months post treatment
  ≥30% improvement in International Prostate Symptom Score (IPSS) score without the need of an additional surgical or minimally invasive procedure. IPSS score ranges from 0-35 (higher score means worse symptoms)
Safety (adverse events) | Within 12 months post treatment
  Frequency and severity of treatment related adverse events will be reported using the Clavien-Dindo severity grading system.

SECONDARY OUTCOMES:
Change in IPSS & IPSS QoL (questionnaire) | 12 months post treatment
  IPSS & IPSS QoL questionnaire
Change in Qmax (maximum flow rate) | 12 months post treatment
  Uroflow to measure maximum flow rate
Change in PVR (post-void residual) | 12 months post treatment
  Bladder scanner to measure post-void residual
Change in sexual function (International Index of Erectile Function, IIEF questionnaire) | 12 months post treatment
  IIEF questionnaire. Lower score in IIEF means worse in erectile dysfunction.
Change in sexual function (Male Sexual Health Questionnaire ejaculatory dysfunction, MSHQ-EjD questionnaire) | 12 months post treatment
  MSHQ-EjD questionnaire. Lower score in MSHQ-EjD means worse in ejaculation function.
Quality of Recovery (QoR) Visual Analogue Scale (VAS) score at 30 days. | 30 days post treatment
  QoR VAS questionnaire. Higher score means good in recovery.
Health care usage | 30 days post treatment
  Procedure time
Health care usage | 30 days post treatment
  Readmission rate within 30days
Rate of repeat surgical intervention | 12 months post treatment
  Number of participants that need repeated surgical intervention

IPD SHARING:
Plan to Share IPD: No